CLINICAL TRIAL: NCT07229924
Title: Effect of Bariatric Surgery on Cognitive Performance Assessed Using a Virtual Reality Program and the Neuropsi Battery.
Brief Title: Evaluation of Cognitive Improvement After Bariatric Surgery Using a Virtual Reality Program and the Neuropsi Neuropsychological Battery
Acronym: CognitiveBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Collaborators: Université de Montréal (Other); NeuroTracker Athletics Inc. (Unknown)
Responsible Party: Principal Investigator, Argelia Pérez Pacheco, Researcher, Hospital General de México Dr. Eduardo Liceaga
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DI/24/501/04/37; DI/24/501/04/37 (Other: Hospital General de México, Dr. Eduardo Liceaga)
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Obesity (Disorder); Obesity and Obesity-related Medical Conditions
Keywords: Bariatric Surgery; Cognition; NeuroTracker; Neuropsi; Obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Evaluation of perceptual-cognitive functions (NeuroTracker) in individuals without obesity.
- Intervention/Treatment (Experimental): Evaluation of perceptual-cognitive functions (NeuroTracker) in patients with morbid obesity or obesity and related conditions, who were treated with bariatric surgery.
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — Surgical procedures designed to induce sustained weight loss in patients with morbid obesity by modifying the gastrointestinal anatomy to restrict caloric intake, reduce nutrient absortion, or alter gut hormonal responses involved in appetite and metabolism regulation.
  Arms: Intervention/Treatment

SUMMARY:
Background: Obesity is a chronic, systemic, and multifactorial disease affecting populations worldwide, with projections indicating a 50% increase by 2035. It is linked to higher risks of cognitive decline, brain atrophy, and neurodegenerative diseases like Alzheimer's. Bariatric surgery has shown benefits in reducing fat and systemic inflammation, which may improve cognitive function. However, the factors predicting such improvements remain unclear.

Objective: To evaluate the effect of bariatric surgery on cognitive performance using virtual reality (Neurotracker) and the Neuropsi neuropsychological battery.

Methods: This prospective quasi-experimental study will include patients with morbid obesity who are candidates for bariatric surgery. Cognitive performance will be evaluated using the Neurotracker virtual reality tool and the Neuropsi neuropsychological battery. Participants will complete Neurotracker sessions three times weekly for two weeks before surgery, and again at 3- and 6-months post-surgery. The Neuropsi assessment will be conducted once prior to surgery and repeated at 6 months afterward. Statistical analyses will compare cognitive performance before and after the surgical intervention.

Expected Outcomes: The study aims to identify measurable improvements in cognitive function after weight loss from bariatric surgery, evaluated through both traditional neuropsychological tests and immersive virtual reality tools. These results could improve understanding of the cognitive benefits of surgical obesity treatment and the factors that predict these outcomes.

ELIGIBILITY:
Inclusion Criteria:

A. Age (18-65 years) B. Diagnostic of morbid obesity with a body mass index (BMI) > 40 kg/m2, or, C. Obesity grade II (BMI > 35 kg/m2) and associated comorbidities (Diabetes Mellitus type 2, Hypertension, Ischemic Cardiopathy, Hyperlipidemia, Hepatic Steatosis, Metabolic Syndrome, Obstructive Sleep Apnea, Pickwick Syndrome) D. Bariatric surgery criteria.

Exclusion Criteria:

A. Age < 18 years, > 65 years B. Visual impairment C. Personal history of CVE D. Drug addiction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
NEUROPSI | NEUROPSI will be applied to group intervention before bariatric surgery and 6 months after it. For the control group, NEUROPSI will be applied at the time of enrollment and 6 months later.
  NEUROPSI is a standardized neuropsychological assessment battery designed to evaluate cognitive functions. It provides quantitative measures adjusted for age and education grade.
NeuroTracker | The time of evaluation will be: 12 sessions pre-surgery, 12 sessions, 3 months post-surgery (post-op) 12 sessions, 6 months post-op With a total of 3 visits per evaluation (9 visits), each patient will complete 80 trials per visit.
  has a virtual cloud-based web portal, that has been validated by functional Magnetic Resonance Imaging. Participants will perform a total of 12 sessions. Each session will consist of 3 blocks of 20 trials.

CONTACTS AND LOCATIONS:
Overall Officials: Argelia Pérez Pacheco, PhD, Principal Investigator — Hospital General de México Dr. Eduardo Liceaga
Locations (2):
- Faubert Lab, Montreal, Quebec, Canada
- Hospital General de México "Dr. Eduardo Licega", Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legault I, Allard R, Faubert J. Healthy older observers show equivalent perceptual-cognitive training benefits to young adults for multiple object tracking. Front Psychol. 2013 Jun 6;4:323. doi: 10.3389/fpsyg.2013.00323. eCollection 2013. PMID 23761025
- [Background] Oria HE, Moorehead MK. Bariatric analysis and reporting outcome system (BAROS). Obes Surg. 1998 Oct;8(5):487-99. doi: 10.1381/096089298765554043. PMID 9819079
- [Background] Hachula M, Kosowski M, Zielanska K, Basiak M, Okopien B. The Impact of Various Methods of Obesity Treatment on the Quality of Life and Mental Health-A Narrative Review. Int J Environ Res Public Health. 2023 Jan 24;20(3):2122. doi: 10.3390/ijerph20032122. PMID 36767489
- [Background] Ostrosky-Solis F, Esther Gomez-Perez M, Matute E, Rosselli M, Ardila A, Pineda D. NEUROPSI ATTENTION AND MEMORY: a neuropsychological test battery in Spanish with norms by age and educational level. Appl Neuropsychol. 2007;14(3):156-70. doi: 10.1080/09084280701508655. PMID 17848126
- [Background] Frigolet ME, Dong-Hoon K, Canizales-Quinteros S, Gutierrez-Aguilar R. Obesity, adipose tissue, and bariatric surgery. Bol Med Hosp Infant Mex. 2020;77(1):3-14. doi: 10.24875/BMHIM.19000115. PMID 32115585
- [Background] Campos-Nonato I, Galvan-Valencia O, Hernandez-Barrera L, Oviedo-Solis C, Barquera S. Prevalencia de obesidad y factores de riesgo asociados en adultos mexicanos: resultados de la Ensanut 2022. Salud Publica Mex. 2023 Jun 14;65:s238-s247. doi: 10.21149/14809. Spanish. PMID 38060949
- See also: Link to the official NeuroTracker website. — https://es.neurotrackerx.com/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT07229924/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT07229924/ICF_001.pdf